CLINICAL TRIAL: NCT04440800
Title: Remote Monitoring of Wearable Activity Trackers for Detection of TOXicity in People Receiving Systemic Anticancer Treatment: a Feasibility Study
Brief Title: Feasibility of Wearable Activity Trackers for Detection of TOXicity in People Receiving Systemic Anticancer Treatment
Acronym: WATTOX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5083
Record Dates: First submitted 2020-02-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer, Small Cell; Pancreatic Cancer; Gastric Cancer; Oesophageal Cancer; Lung Cancer, Nonsmall Cell; Lung Cancer Metastatic
MeSH Terms: conditions — Small Cell Lung Carcinoma; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study participants: All patients will receive the intervention
  Interventions: Device: Wearable activity tracker - FitBit

INTERVENTIONS:
Device: Wearable activity tracker - FitBit — Participants will be given a wearable activity tracker and their daily step count recorded. If there is a reduction from baseline of over 1000 steps, the participant will be contacted and an ambulatory review organised if the reduction is not due to a device compliance issue

SUMMARY:
Accurate evaluation of activity status is an important part of the assessment of people with cancer. Clinician assessments currently used are valuable but have limitations; in particular, assessment only occurs when the patient attends clinic and is often subjective. Activity trackers, such as FitBits, give the opportunity to objectively assess activity status continuously, independent of clinic visits. Previous studies have shown that a reduction in 1000 steps while receiving cancer treatment is associated with an increased risk of hospitalisation but it is not known if using information from activity trackers to allow early intervention is feasible or if it can reduce admission to hospital and improve outcomes.

The investigators propose a prospective feasibility study in people with advanced lung cancer or upper gastrointestinal cancers who are starting a new line of systemic anti-cancer therapy.

Participants will receive a FitBit, which is a commercially available wearable activity tracker for the duration of their treatment or 4 months (whichever is shorter). Step counts will be monitored and a reduction in daily steps of >1000 from baseline will trigger contact by the study team and an ambulatory review. Participants will not receive treatment within the context of the study.

DETAILED DESCRIPTION:
A recent metanalysis reports that over 40% of people with cancer being treated with palliative intent have at least 1 unplanned hospital admission during treatment. Furthermore, up to 83% of people undergoing cancer treatment are likely to attend the Emergency Departments (ED). The 2019 NHS long-term plan has an emphasis on the use of digital technologies, remote monitoring to support patients, and acute ambulatory care as an alternative to ED attendance.

In observational studies of people with cancer, reductions in steps counts correlate with increased symptoms and risk of hospitalisation.

Therefore, the main aim of this study is to determine whether monitoring of activity and subsequent ambulatory review triggered by detecting a reduction in steps is feasible in a timely fashion within an NHS oncology centre.

People with advanced lung cancer (NSCLC, SCLC) or upper gastrointestinal cancers (gastric, oesophageal or pancreatic) starting a new line of systemic anti-cancer treatment (SACT) will be recruited at The Royal Marsden Hospital (Chelsea and Sutton sites). Eligible patients will be approached by clinical teams in the lung and gastrointestinal cancer outpatient clinics.

Participants who are due to start a new line of SACT will be asked to wear a FitBit activity tracker (resembling a watch). Baseline median daily steps count will be calculated prior starting SACT for those patients who wear the device for ideally 7 consecutive days, which must include both weekend and week days.

The device can measure step counts and heart rate. The FitBit will be monitored remotely by the study team once a day (week days only) using a web-based platform called Fitabase and will document cases where the step count reduction is >1000 from baseline. Step count and average heart rate data will be downloaded at the beginning of each treatment cycle and a summary reported in the MACRO database. Fitabase is a cloud-based data management platform, which is able to access data which has been synchronised from individual FitBits. Data can be collected anonymously by associating the device data with a study identification number. Fitabase does not collect personally identifiable data. No global positioning system (GPS) data or other data is collected. Passwords are encrypted.

For this feasibility study, activity tracking will take place on working week days only.

A reduction in >1000 steps from the baseline median step count will trigger a telephone call by a member of the study team. If the fall in steps was not due to non-compliance/malfunction of the device, the participant will be invited to attend the Clinical Assessment Unit for an ambulatory review. Participants' acceptance of advice to attend for a review will be documented. The diagnosis (and clinical necessity as assessed by a clinician), need for hospitalisation or not, and length of stay will be collected. Further investigations or management will be determined by clinical need following assessment by a member of the study team.

If no abnormality is noted the trigger for subsequent phone calls will be adjusted by 500 steps for that patient ie >1500 steps. If no abnormality is found after a second review, further reviews will only take place after a phone call if there is clinical concern.

Participants will be informed at the beginning of the study to use usual processes if they feel unwell at any time eg calling the Royal Marsden Macmillan Hotline (RMMH).

Participants will be reviewed at the start of each new cycle of treatment (+/- 7 days) by a member of the study team to find out if they have been hospitalised and for how long.

Physician-assessed PS, C reactive protein (CRP), albumin, handgrip strength (HGS), Timed Up and Go (TUaG) will be measured at the first study visit, and skeletal muscle area (SMA), skeletal muscle index (SMI) and muscle radiation attenuation (MRA) will be measured from the standard of care baseline CT scan. In addition the investigators will also collect height and weight demographics, and perform questionnaire-based nutritional (PG-SGA) and quality of life (QoL) (FACT-G, EORTC-q30C) assessments.

To assess changes in muscle quality and function, HGS, PS, and TUaG will be measured +/- 14 days from each standard of care CT scan. The participant will also undertake QoL and nutrition questionnaires as per baseline investigation. Weight will be recorded. The CT scan will be used to calculate SMA, SMI and MRA.

At the end of the study, 5-8 participants will be invited for a focus group to understand their acceptance and experience of remote activity monitoring while undertaking cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18.
* Advanced lung (NSCLC or SCLC) cancer or patients with upper gastrointestinal cancer (gastric, oesophageal, pancreatic) starting a new line of systemic anti-cancer therapy.
* Willingness to wear an activity tracker and undergo remote monitoring
* Access to a smart phone.
* Willingness to have a Fitbit App installed on their smartphone
* Willingness to have a pseudo- anonymised FitBit account created for the purposes of the study
* PS 0-2.
* 1 or more previous lines of treatment.

Exclusion Criteria:

* Physical conditions that preclude daily walking
* Inability to give informed consent.
* Medical or psychiatric condition which in the investigators opinion would affect the successful completion of the study.
* Immediate need to start systemic anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant population whose data will be subjected to the study analysis includes registered patients for whom baseline median daily step count was available and who were compliant with wearing the device during the follow up.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of monitoring reductions in step count in people with advanced lung cancer or upper gastrointestinal cancers starting systemic anti-cancer therapy. | Analysis 4 months after last patient recruited
  Feasibility of step count monitoring will be determined by measuring the proportion of participants for whom step count was successfully monitored (step count checked for at least 4 out 5 weekdays) for at least 80% of the treatment weeks during the study period.
  Successful monitoring is defined as a member of the study team logging in to the Fitabase system to review the step count. If 80% of participants are monitored for 80% of the observational time (from the start until the end of treatment - either at completion or if treatment is stopped), this will be considered feasible.
Feasibility of undertaking a timely ambulatory review, of participants in whom a reduction of steps is detected | Analysis 4 months after last patient recruited
  Feasibility of a timely ambulatory review will be determined by measuring the proportion of participants who are invited for an ambulatory review and attend within 24 hours. If 70% of participants invited for a review attend, this will be considered feasible.

SECONDARY OUTCOMES:
Participant compliance with use of activity monitor | Analysis 4 months after last patient recruited
  Percentage compliance with wearable activity trackers (WAT) will be defined as wearing the device for at least 70% of waking hours. It is assumed for the purposes of this study that participants are awake between 0700hrs to 2200hrs. Compliance can be assumed if the device is able to measure heart rate during these hours, which can be assessed from the daily heart rate graph.
Utility of monitoring steps counts as a trigger for ambulatory assessment for the identification of new or worsening adverse events in people with cancer. | Analysis 4 months after last patient recruited
  The utility of monitoring steps counts for the identification of new or worsening adverse events in people with cancer will be assessed by recording the number of clinical reviews triggered by step count.
Sensitivity of monitoring steps counts for the identification of new or worsening adverse events in people with cancer | Analysis 4 months after last patient recruited
  The sensitivity of monitoring steps counts for the identification of new or worsening adverse events in people with cancer will be assessed by recording how many of the triggered ambulatory assessments were deemed clinically appropriated by the assessing clinician.
Number of hospitalisation episodes. | Analysis 4 months after last patient recruited
  The total number of hospitalisation episodes will be recorded, including all WAT-triggered ambulatory reviews and those that occur outside of the study visits
Proportion of hospitalisation episodes associated with WAT-triggered ambulatory reviews. | Analysis 4 months after last patient recruited
  The proportion of hospitalisation episodes that were WAT-triggered clinical reviews, including those with no detected abnormality, will be compared to the number of episodes that were not associated with a WAT-triggered review.
Acceptability of remote activity tracking | At study completion, approximately 1 year after beginning recruitment
  Acceptability of remote activity tracking will be determined by assessing the qualitative patient experience of undergoing remote monitoring as determined by focus group interview

OTHER OUTCOMES:
Correlation between steps count, physician assessed WHO performance status (PS), quality of life (QoL) and muscle mass/attenuation/function | Analysis 4 months after last patient recruited
  To explore the correlation between /median step-count and:
  1. physician assessed PS as recorded at treatment visits or CT
  2. SMA, SMI and MRA
  3. HGS
  4. TUaG
  5. QoL (as assessed by FACT-G and EORTC-q30C).
  6. Nutrition (as assessed by BMI and PG-SGA)
Correlation between resting heart rate, hospitalisation and muscle mass/attenuation/function | Analysis 4 months after last patient recruited
  To explore the correlation between changes in resting heart rate from baseline and mean/median steps, hospitalisation, HGS, SMA, SMI and MRA

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Yousaf, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - London and Surrey, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohri N, Kabarriti R, Bodner WR, Mehta KJ, Shankar V, Halmos B, Haigentz M Jr, Rapkin B, Guha C, Kalnicki S, Garg M. Continuous Activity Monitoring During Concurrent Chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2017 Apr 1;97(5):1061-1065. doi: 10.1016/j.ijrobp.2016.12.030. Epub 2016 Dec 25. PMID 28332990
- [Background] Gresham G, Hendifar AE, Spiegel B, Neeman E, Tuli R, Rimel BJ, Figlin RA, Meinert CL, Piantadosi S, Shinde AM. Wearable activity monitors to assess performance status and predict clinical outcomes in advanced cancer patients. NPJ Digit Med. 2018 Jul 5;1:27. doi: 10.1038/s41746-018-0032-6. eCollection 2018. PMID 31304309
- [Background] Prince RM, Powis M, Zer A, Atenafu EG, Krzyzanowska MK. Hospitalisations and emergency department visits in cancer patients receiving systemic therapy: Systematic review and meta-analysis. Eur J Cancer Care (Engl). 2019 Jan;28(1):e12909. doi: 10.1111/ecc.12909. Epub 2018 Sep 20. PMID 30238542
- [Background] Bennett AV, Reeve BB, Basch EM, Mitchell SA, Meeneghan M, Battaglini CL, Smith-Ryan AE, Phillips B, Shea TC, Wood WA. Evaluation of pedometry as a patient-centered outcome in patients undergoing hematopoietic cell transplant (HCT): a comparison of pedometry and patient reports of symptoms, health, and quality of life. Qual Life Res. 2016 Mar;25(3):535-46. doi: 10.1007/s11136-015-1179-0. Epub 2015 Nov 17. PMID 26577763
- [Background] Spruit MA, Sillen MJ, Groenen MT, Wouters EF, Franssen FM. New normative values for handgrip strength: results from the UK Biobank. J Am Med Dir Assoc. 2013 Oct;14(10):775.e5-11. doi: 10.1016/j.jamda.2013.06.013. Epub 2013 Aug 16. PMID 23958225
- See also: NHS England. NHS Long Term Plan January 2019 — https://longtermplan.nhs.uk/online-version